CLINICAL TRIAL: NCT02683694
Title: Characteristics and Limitations of Intraoperative OCT Supported Membrane Peeling in Macular Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim. Prof. Dr. Oliver Findl, MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iOC
Record Dates: First submitted 2016-02-12; First posted 2016-02-17 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Macular Diseases
Keywords: Epiretinal membrane; lamellar holes of the macula; macular holes; vitreomacular traction syndrome
MeSH Terms: conditions — Epiretinal Membrane; Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- study arm (Other): iOCT is performed
  Interventions: Device: iOCT

INTERVENTIONS:
Device: iOCT — the number of subjects that can be peeled without dye are assessed
  Other Names: intraoperative OCT (iOCT)

SUMMARY:
During the last decade optical coherence tomography (OCT) extended the possibilities for in vivo macula diagnostic and was increasingly used for pre- and post-operative imaging of retinal diseases. Spectral-domain optical coherence tomography (SD-OCT) with its increased scanning speed and image-resolution provides more detailed information of microstructures in the macula.

Epiretinal membrane (ERM), lamellar macular hole, macular hole and vitreomacular traction syndrome are disorders involving the posterior pole of the eyeball with consecutive vision loss. In patients with loss of vision and metamorphopsia disturbing their lifestyle, vitrectomy and membrane peeling is usually performed to remove traction and the ERM.

Different study groups showed that intraoperative use of SD-OCT is possible and improves the quality of peeling surgery.

DETAILED DESCRIPTION:
The aim of the study is to assess the benefits and limits of intraoperative OCT (i-OCT), for example whether I-OCT assisted membrane peeling is possible without use of dyes for enabling better localistion of the ERM during surgery and to compare that scheme with different "gold standard" dyes for peeling such as membrane blue dual and triamcinolone. Rationale for that study is to work out which setting enables best visualisation of ERM and ILM (ILM) in i-OCT. A limitation of that method seems to be visualisation of the inner limiting membrane, so that dying of the ILM will probably be still necessary in all cases where ILM-peeling is sheduled.

ELIGIBILITY:
Inclusion Criteria:

* Epiretinal Membrane, lamellar hole of the macula, macular hole and vitreomacular traction syndrome

Exclusion Criteria:

* Other diseases of the eye, such as AMD, retinopathia pigmentosa

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-02; Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
peeling without staining | intraoperative (10-15 minutes)
  number of patients that could be peeled without use of a dye

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- VIROS, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided